CLINICAL TRIAL: NCT06347575
Title: Safety and Tolerability of a Novel Implantable Neurostimulator for Ameliorate Erectile Function: a Pilot Study in Spinal Cord Injured Patients
Brief Title: Safety and Tolerability of a Novel Implantable Neurostimulator for Ameliorate Erectile Function on Spinal Cord Injured Patients
Acronym: CAVERSTIM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The company that supplies the Medical Device has withdrawn.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Comphya SA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP230522
Record Dates: First submitted 2023-10-02; First posted 2024-04-04 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injuries; Erectile Dysfunction
Keywords: spinal cord injuried; penile erection; electrical stimulation; implantable; pilot study; cavernous nerve
MeSH Terms: conditions — Spinal Cord Injuries; Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantation of the caverStim device (Experimental): Implantation of caverStim in SCI patients
  Interventions: Device: Implantation of the caverStim device

INTERVENTIONS:
Device: Implantation of the caverStim device — Implantation of caverStim in SCI patients.

SUMMARY:
The main objective of the study is to assess the safety and tolerability of cavernous nerve electrical stimulation in patients with spinal cord injured (SCI) by assessing and measuring complications.

As the secondary objectives, despite the limited cohort size, this long-term study aims to obtain preliminary data on efficacy of cavernous nerve stimulation to improve erectile function for sexual intercourse, as well as to assess patient's satisfaction using:

* Objective assessment of the erectile response upon CaverSTIM activation with the RigiScan device.
* Subjective assessment of the erectile function with validated questionnaires:

  1. A 6-item self-report instrument assessing male erectile function (Erectile Function domain of the International Index of Erectile Function, IIEF-EF);
  2. A log-diary five item questionnaire completed after each sexual attempt (Sexual Encounter Profile, SEP);
  3. A self-reporting measure that scores erection hardness on a 4-point scale (Erection Hardness Score, EHS);
  4. The Global Assessment Question (GAQ).

In addition, the study aims to refine the method of implantation (step-by-step delineation of all technical approaches for device implantation, including duration of surgical procedure, blood loss, methods to access the periprostatic region, tissue dissection, device placement and fixation) prior to planning for larger scale clinical investigation.

DETAILED DESCRIPTION:
Depending on the location and whether the spinal cord lesion is complete or not, oral medications (phosphodiesterase type 5 (PDE5-Is) inhibitors, eg Viagra®) may be more or less effective in improving erectile function. When these drugs are not sufficiently effective, the second-line pharmacological treatment for SCI patients consists of intracavernous injections. Treatment by intracavernous injections is responsible for additional constraints. Indeed, a titration must be carried out in a doctor's office (important to minimize the risk of priapism). Specific learning of the injection technique must also be implemented for the patient and/or his partner, the identification of the injection site (laterally in the cavernous bodies at an angle of 90° with respect to the long axis of penis, avoiding the urethra and subcutaneous veins) and aseptic handling. The use of intracavernous injections is often abandoned by patients due to a high level of discomfort, complicated self-injection or lack of spontaneity during sexual intercourse. In patients with SCI, intracavernous injections of prostaglandin E1 fail to induce a sufficiently rigid erection in 20% of them. Vacuum device is another option. Nevertheless it may be perceived as cumbersome and lacking of spontaneity. In case of failure or lack of acceptance of intracavernous injections and vacuumdevice, the penile implant, which consists of a pair of malleable or inflatable cylinders surgically implanted in the cavernous bodies previously destroyed surgically, is the third-line treatment. However, penile implants have an increased risk of infection in patients with SCI, according to two large studies. Thus, effective, acceptable and safe treatment alternatives are sought by patients with SCI who are insufficiently responsive to oral treatments.

The concept of electro-neurostimulation therapy to activate the cavernous nerves for erectile dysfunction was introduced two decades ago. Despite its recognized potential and the first promising studies confirming the feasibility of peri-prostatic cavernous nerve stimulation, this technology has not yet been developed. The difficulty lies in the complex anatomy of the human cavernous nerve. Indeed, it is difficult to identify the optimal site for stimulation because the human cavernous nerve is not visible on a macroscopic scale and extends from the pelvic plexus to the penis through a peri-vesical and peri-prostatic neuroplexus. whose anatomy is complex. In addition, the course of the cavernous nerve is subject to strong interindividual variability. In addition to these intrinsic anatomical problems, other difficulties are encountered during the surgical intervention, such as the presence of overlying tissues, connective tissue and potential bleeding obstructing the operative field, thus making the optimal placement of the implants complex.. The main difficulty in applying neurostimulation to the treatment of erectile dysfunction is therefore to identify the stimulation site to place the stimulation electrodes in optimal contact with the cavernous nerve.

A practical solution was invented by a patch with twelve electrodes. This solution was designed to promote extensive contact with the cavernous nerve. The concept was developed to allow implantation of the electrodes regardless of the visibility of the cavernous nerve bundles. This concept makes it possible to globally cover the anatomical region of interest where the cavernous nerve is supposed to be located, while taking into account the great heterogeneity of its course. This approach then guarantees optimal contact of at least a few electrodes with the cavernous nerve and thus offers optimal stimulation conditions.

The multi-electrode patches will be implanted during a robotic laparoscopic surgical procedure. A stimulation test will be performed during the operation to ensure that the patient responds to stimulation (erectile response) before the device is permanently implanted. Following the recovery of the patient, the selection of the stimulation parameters will be carried out on an outpatient basis in order to identify the electrode(s) which give(s) the best erectile response. The electrodes in contact with the cavernous nerve bundles (causing the maximum erectile response) will then be selected and recorded for stimulation/therapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects have to fulfill all of the following inclusion criteria before being included in the run-in phase:

* Written informed consent obtained from the subject;
* Men between the age of 18 to 45 years old with supra sacral spinal cord injury and below T6 as the upper limit;
* Men with stable spinal cord injury, which occurred at least 6 months prior to study enrolment;
* Men with documented neurogenic overactive detrusor activity according to urodynamic testing in their files;
* Have a monogamous relationship with a female sexual partner (vaginal penetration required for several of the primary efficacy variables) for at least 6 months prior to screening
* Men with an insufficient response to PDE5-Is and interested in treating erectile dysfunction;
* Ability to understand and follow study-related instructions.

Subjects have to fulfill all of the following inclusion criteria before being included in the implantation phase:

* At least 4 sexual intercourse attempts during the 4-week run-in phase with use of 100 mg sildenafil approximately 1 hour before attempting intercourse
* IIEF-EF score < 17 at the end of the run-in phase;
* At least 50% of attempts at sexual intercourse during the run-in phase had been unsuccessful i.e. the following question in the SEP Diary had to be answered with "No":

"Did your erection last long enough for you to have successful intercourse?" (SEP3: success in maintenance of erection).

Exclusion Criteria:

All exclusion criteria will be assessed before the 4-week run-in phase.

The presence of any one of the following exclusion criteria will lead to exclusion of the subject:

* Patients with spinal cord lesion at T6 or above;
* Patients with known allergies to any of the device material (Platinum/iridium, silicone, pellethane, titanium, polysulfone, polyurethane);
* Patients contraindicated for surgery under general anesthesia;
* History of priapism or Lapeyronie's disease;
* Patients having met the criteria for unstable angina within 6 months prior to Visit 1, history of myocardial infarction or coronary artery bypass graft surgery within 90 days prior to Visit 1, or percutaneous coronary intervention (eg, angioplasty or stent placement) within 90 days prior to Visit 1.
* Any supraventricular arrhythmia with an uncontrolled ventricular response (mean heart rate >100 bpm) at rest despite medical therapy, or any history of spontaneous or induced sustained ventricular tachycardia (heart rate >100 bpm for >=30 sec) despite medical therapy;
* A history of sudden cardiac death (arrest) despite medical therapy.
* Any evidence of congestive heart failure within 6 months prior to Visit 1.
* History of previous pelvic surgery or irradiation therapy;
* Prior surgery for an implantable penile prosthesis;
* Inability to understand and to follow instructions on device use;
* Patients with diabetes mellitus
* Patients not interested in sexual activity;
* Patients currently participating in another clinical investigation;
* Patient has participated in any drug or device trial in the last 4 weeks or plans to participate in any other drug or device study in the next 24 months;
* Any other characteristics that, per the investigator's judgment, may increase the patients risk or impair the study conduct and data collection; such as depression or abnormal behavior for example.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | at 6 months
  The safety of the CaverSTIM device will be assessed by systematically reporting device failures, adverse events including serious adverse events, while monitoring the frequency, severity and incidence of these events.
Pain assessement | at 6 months
  Pain will be assessed during the days following the implant surgery as well as during activation of the device, by asking the subject to rate their pain from 0 to 10 using a visual analogue scale (VAS).
Complications related to implantation surgery | at 6 months
  Complications related to implantation surgery should be evaluated and classified according to the Clavien-Dindo classification.

SECONDARY OUTCOMES:
Evaluation of IIEF-EF | at 6 months
  Subjective evaluation of penile erection and sexual satisfaction of the subject by means of validated questionnaires:
  IIEF-EF (Erectile Function domain score from the International Index of Erectile Function)
Evaluation of EHS | at 6 months
  Subjective evaluation of penile erection and sexual satisfaction of the subject by means of validated questionnaires:
  EHS (Erection Hardness Score)
Evaluation of SEP | at 6 months
  Subjective evaluation of penile erection and sexual satisfaction of the subject by means of validated questionnaires:
  SEP (Sexual Encounter Profile)
Evaluation of GAQ | at 6 months
  Subjective evaluation of penile erection and sexual satisfaction of the subject by means of validated questionnaires:
  GAQ (Global Assessment Question).

CONTACTS AND LOCATIONS:
Overall Officials: François Giuliano, MD, PhD, Principal Investigator — Department of neurology-urology-andrology, Raymond Poincaré hospital - APHP; Emmanuel CHARTIER-KASTLER, MD, PhD, Study Director — Department of Urology, La Pitié-Salpétrière hospital - APHP; Anne Charlotte DENORMANDIE, MD, Study Director — Department of Urology, La Pitié-Salpétrière hospital - APHP
Locations (1):
- Department of neurology-urology-andrology, Raymond Poincaré hospital - APHP, Garches, France